CLINICAL TRIAL: NCT01402401
Title: An Open-label, Single-arm, Multi-center Phase II Study to Evaluate the Efficacy and Safety of AUY922 in Combination With Trastuzumab Standard Therapy as Second-line Treatment in Patients With HER2-positive Advanced Gastric Cancer
Brief Title: Phase II of AUY922 in Second-line Gastric Cancer in Combination With Trastuzumab in HER2 Positive Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2205; 2011-002570-23 (EudraCT Number)
Record Dates: First submitted 2011-07-24; First posted 2011-07-26 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-08

CONDITIONS: Advanced Gastric Cancer
Keywords: HER2+,; Gastric Cancer,; HSP90,; 2nd-line,; Trastuzumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Trastuzumab

ARMS (1):
- AUY922 + Trastuzumab (Experimental)
  Interventions: Drug: AUY922; Drug: Trastuzumab

INTERVENTIONS:
Drug: AUY922
Drug: Trastuzumab

SUMMARY:
This study will assess the safety and efficacy of AUY922, when administered, in combination with trastuzumab in adult patients with HER2+ advanced gastric cancer, who have received trastuzumab plus chemotherapy in the first line.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

1. Written informed consent obtained prior to any screening procedures
2. Patients with documented cytological or histological confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma and proven HER2 positive.
3. Patients with progressive disease (radiological confirmation required according to RECIST) after first line of trastuzumab in combination with chemotherapy for advanced gastric cancer.
4. Age ≥ 18 years or age of consent in country of residence and able to sign Informed Consent
5. ECOG performance status of 0-1 at study entry
6. HER2-overexpressing positive gastric tumor by IHC3+ or IHC2+ with positive in situ hybridization
7. Measurable disease according to RECIST (Irradiated lesions can not be considered measurable unless they have clearly progressed since radiotherapy).
8. Negative serum pregnancy test. The serum pregnancy test must be obtained prior to any drug administration (≤ 72 hours prior to dosing) in all pre-menopausal women and for women < 2 years after the onset of menopause.
9. Patients must have the following laboratory values:

Hematologic

* Absolute Neutrophil Count (ANC) ≥1.5x109/L,
* Hemoglobin (Hgb) ≥ 9 g/dL,
* Platelets (plt) ≥100x109/L

Biochemistry:

* Serum total bilirubin ≤ 1.5 x ULN
* Serum albumin > 2.5 g/dl
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 ml/min.
* AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

1. Evidence of spinal cord compression or current evidence of CNS metastases. CT/MRI of the brain is mandatory (within 3 weeks before study start) in case of clinical suspicion or evidence of brain metastases
2. Patient who are < 4 weeks since last chemotherapy or treatment with another systemic anti-cancer agent. Patients must have recovered (CTC ≤ 1) from acute toxicities of any previous therapy (with the exception of alopecia).
3. Patients may have received prior radiotherapy for management of local disease providing that disease progression has been documented, all toxicities have resolved (CTC ≤ 1) (with the exception of alopecia), and the last fraction of radiotherapy was completed at least 4 weeks prior to the study.
4. Prior treatment with an agent that acts via HER2/c-erbB2 targeting other than 1st line trastuzumab, include (but are not limited to) lapatinib and pertuzumab.
5. Treatment with therapeutic doses of coumarin-type anticoagulants. (Maximum daily dose of 2 mg, for line patency permitted)
6. Patients with malignant ascites that require invasive treatment
7. Patients with acute or chronic renal disease; and active and chronic liver disease requiring intervention. Other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol.
8. Major surgery ≤ 2 weeks prior to enrollment or who have not recovered from such therapy
9. Impaired cardiac function
10. Concurrent malignancies or invasive cancers diagnosed within the past 5 years, except for adequately treated basal cell cancer of the skin or in situ cancer of the cervix
11. Patients receiving chronic or high dose corticosteroids therapy (Inhaled steroids and short courses of oral steroids for anti-emesis or as an appetite stimulant are allowed)
12. Patients unwilling or unable to comply with the protocol
13. Patients known to be HIV positive. Testing is not required in the absence of clinical signs and symptoms suggesting HIV infection.
14. Known hypersensitivity to any of the study drugs or their excipients
15. Participation in another clinical study within 30 days before first study treatment
16. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
17. Fertile women of childbearing potential (WOCBP) not using adequate contraception (abstinence, oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
efficacy of AUY922 in combination with trastuzumab as assessed by RECIST | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United States (3):
  - University of California at Los Angeles UCLA LeConte Location, Los Angeles, California
  - Clinical Research Alliance, Lake Success, New York
  - University of Texas/MD Anderson Cancer Center UT SC, Houston, Texas
- Novartis Investigative Site, Leuven, Belgium
- France (3):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Reims
- Germany (2):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Heilbronn
- Novartis Investigative Site, Modena, MO, Italy
- Japan (2):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- See also: Results for CAUY922A2205 can be found on the Novartis Clinical Trial Results website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=11163